CLINICAL TRIAL: NCT03260465
Title: A Randomized Controlled Trial With the seleXys PC Cup and RM Pressfit Vitamys Cup in Combination With the Optimys Short Stem
Brief Title: Clinical Study With the seleXys PC and the RM Pressfit Vitamys Cup
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-00832; mu21Stoffel
Record Dates: First submitted 2017-08-22; First posted 2017-08-24 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Hip Joint; Arthritis, Degenerative
Keywords: total hip replacement; roentgen stereophotogrammetric analysis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Intervention Model Description: prospective, randomised single-center study with 2 treatment arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- seleXys PC (Experimental): seleXys PC cup combined with the optimys stem
  Interventions: Device: seleXys PC
- RM (Active Comparator): RM Pressfit vitamys cup combined with the optimys stem
  Interventions: Device: RM

INTERVENTIONS:
Device: seleXys PC — Total hip arthroplasty using the seleXys PC cup
  Arms: seleXys PC
Device: RM — Total hip arthroplasty using the RM cup
  Arms: RM

SUMMARY:
This is a randomized controlled trial with the seleXys PC cup and RM Pressfit vitamys cup in combination with the optimys short stem. Wear rate and migration is assessed with roentgen stereophotogrammetric analysis (RSA) measurements.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic arthritis who are candidates for a primary total hip arthroplasty with an uncemented femoral stem as determined jointly by the surgeon and the patient.
* Patients suitable for an uncemented acetabular component in combination with a 36mm femoral head (seleXys PC cup: 52mm, 54mm or 56mm; RM Pressfit vitamys: 52mm, 54mm or 56mm)
* Patients between the ages of 50 and 75 inclusive
* Patients who understand the conditions of the study and are willing to participate for the length of the prescribed follow-up

Exclusion Criteria:

* Patients that require an acetabular cup size which cannot be used in combination with a 36mm femoral head
* Patients that offer no guarantee for regular follow-up controls
* Patients that have a revision surgery
* Patients that have a fracture of the femoral neck or a bone tumour in the area of the femur or pelvis
* Patients that had a previous osteotomy of the femur or pelvis
* Pregnant women or those seeking to become pregnant
* Patients with a history of active infection

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Wear Rate | 3 years
  The principal purpose of this study is to compare the modular seleXys PC Cup with a vitamys inlay to the monoblock RM Pressfit vitamys cup by means of wear rate. In addition, the migration of the two cups and the optimys stem, respectively, will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Karl Stoffel, Prof. Dr. med., Principal Investigator — Klinik für Orthopädie und Traumatologie, Universitätsspital Basel
Locations (1):
- Klinik für Orthopädie und Traumatologie, University Hospital Basel, Basel, Basel-Landschaft, Switzerland

IPD SHARING:
Plan to Share IPD: No